CLINICAL TRIAL: NCT02401750
Title: A Multi-center, Randomized, Multiple-dose, Double-blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Abuse-deterrent Capsules Oxycodone Hydrochloride Plus Naltrexone Hydrochloride (a) or Oxycodone Hydrochloride Plus Naltrexone Hydrochloride (b) for the Treatment of Adults With Moderate to Severe Pain Following Bunionectomy Surgery
Brief Title: A Study to Evaluate Safety and Efficacy Following Dosing of Oxycodone/Naltrexone for Treatment of Adults With Pain Following Bunionectomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elite Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELI-003-2014
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxycodone Naltrexone (a) (Experimental): Double-Blind Oxycodone/Naltrexone, 1 capsule by mouth every 6 hours for 48 hours
  Interventions: Drug: Oxycodone Naltrexone (a)
- Oxycodone Naltrexone (b) (Experimental): Double-Blind Oxycodone/Naltrexone , 1 capsule by mouth every 6 hours for 48 hours
  Interventions: Drug: Oxycodone Naltrexone (b)
- Placebo (Placebo Comparator): Double-Blind Placebo to experimental Oxycodone/Naltrexone, 1 capsule every 6 hours for 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone Naltrexone (a)
  Arms: Oxycodone Naltrexone (a)
Drug: Oxycodone Naltrexone (b)
  Arms: Oxycodone Naltrexone (b)
Drug: Placebo — Matches both experimental drugs
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, Phase 3 study to evaluate the efficacy and safety of the administration of multiple doses of Oxycodone Hydrochloride plus Naltrexone Hydrochloride (a) or Oxycodone Hydrochloride plus Naltrexone Hydrochloride (b) in patients who have undergone primary, unilateral, distal first metatarsal bunionectomy with osteotomy and internal fixation.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety and efficacy of oxycodone/naltrexone (a) and oxycodone/naltrexone (b) versus placebo. During the blinded phase of the study (inpatient portion) the dosing regimen is 1 capsule containing Oxycodone Hydrochloride plus Naltrexone Hydrochloride (a) or Oxycodone plus Naltrexone Hydrochloride (b) or placebo taken with 4 to 6 ounces (oz) of water every 6 hours (q6h) for 48 hours following the first dose (Multiple-dose Period) while in-house. Then for the open-label phase of the study (outpatient portion) dosing will occur every 4 to 6 hours prn with Oxycodone plus naltrexone. The active and placebo study medications will appear identical. Study subjects with acute postoperative pain of moderate to severe intensity following unilateral bunionectomy surgery will be randomized after surgery, and will stay at the study center for the duration of the 48-hour double-blind period after dose 1 of study medication. The study will be conducted in the following 4 periods: 1) a pre-treatment period, 2) a multiple-dose inpatient period (double-blind), 3) a multiple-dose outpatient period (open-label), and 4) End of Study/Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Complete the informed consent process as documented by a signed informed consent form (ICF).
2. Be in generally good health and classified as either PS-1 or PS-2 by the American Society of Anesthetists (ASA) Physical Status Classification System.
3. Be male or female, age 18 to 75 years, inclusively at the time of screening.
4. Be scheduled for a primary, unilateral, distal, first metatarsal bunionectomy with osteotomy and internal fixation (with no collateral procedures)
5. Female subjects are eligible only if all of the following apply:

   * Not pregnant (subjects of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (B-hCG) pregnancy test at screening and a negative urine pregnancy test before surgery);
   * Not lactating;
   * Not planning to become pregnant within the duration of study;
   * Surgically sterile (bilateral tubal ligation or hysterectomy), or at least two years postmenopausal, or is practicing an acceptable form of birth control (defined as the use of an intrauterine device [IUD], a barrier method with spermicide, condoms, any form of hormonal contraceptives, partner with a vasectomy (surgery at least 6 weeks prior to start of surgery) or abstinence ) for at least 3 months prior to the screening visit and agrees to continue acceptable methods of contraception until one week following the last dose of ELI-200.
6. Be willing to complete the pain assessments and return to clinic as scheduled.
7. Subjects must experience postoperative pain (Day 1) that is at least moderate as measured by a NRS score ≥ 4 on a 0-10 NRS, less than 9 hours after discontinuing the nerve block.

Exclusion Criteria:

1. Have an uncontrolled medical condition, serious intercurrent illness, clinically significant general health condition, or extenuating circumstance that may significantly decrease study compliance or otherwise preclude their participation in the study.
2. Have a clinically significant abnormal electrocardiogram (ECG) at screening as determined by the Investigator.
3. Have had any type of gastric bypass surgery or have a gastric band. Have previous abdominal surgery within the past year or history of abdominal adhesions, known or suspected paralytic ileus.
4. Have a history of any medical condition or surgical procedure that would alter the absorption, distribution, metabolism or excretion of oxycodone or any opioid including but not limited to severe chronic diarrhea, chronic constipation, irritable bowel syndrome, or bowel resection.
5. Have a history of severe bronchial asthma, hypercarbia, or hypoxia (oxygen partial pressure [PO2] <92%) or any respiratory condition that, in the opinion of the investigator, makes the subject unsuitable for the study. Mild episodic asthma or exercised induced asthma will be allowed.
6. Have, in the opinion of the investigator, a clinically significant abnormality on their clinical laboratory values (urinalysis, hematology and chemistry) at screening.
7. Have glycosylated hemoglobin (2c) > 7%.
8. Have Addison's disease, benign prostatic hyperplasia, or kidney disease or other conditions as outlined in the Investigator's Brochure or the Percocet and Oxycontin Package Inserts that are contraindicated for use.
9. Have made a donation (standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 56 days prior to Day -1 .
10. Have made a plasma donation within 7 days prior to Day -1.
11. Have a known allergy or hypersensitivity to any opioid analgesics, naltrexone, anesthetics (eg, propofol), acetaminophen, NSAIDs (eg, ibuprofen or naproxen, ketorolac) or any of the excipients
12. Have a known allergy or hypersensitivity to ropivacaine, Mepivacaine, Lidocaine or any related drug.
13. Have a history of significant intolerance (in the opinion of the investigator) or allergic hypersensitivity reaction to opioid use.
14. Not be willing to discontinue the prohibited medications, within the allotted time before surgery and throughout the duration of their participation in the study.
15. Have a history of substance(more than recreational use) or alcohol (more than 14 drinks in a week) abuse within 2 years before screening.
16. Have a positive drug screen or alcohol screen result.
17. Use of anti-coagulant agents (eg, Coumadin, heparin, etc)
18. Have a positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at the screening visit.
19. Have an active malignancy of any type, or has been diagnosed with cancer within 5 years prior to screening (excluding squamous or basal cell carcinoma of the skin).
20. Have dysphagia and/or cannot swallow study medication whole.
21. Use concurrent therapy that could interfere with the evaluation of efficacy or safety parameters in the opinion of the investigator. (eg, any drugs, in the investigators opinion, that may exert significant analgesic properties or act synergistically with oxycodone, morphine, ketorolac, acetaminophen or ibuprofen).
22. Have a history of seizures or history of serious head injury.
23. Must not be a member of a vulnerable population as defined by the Code of Federal Regulations Title 45, Part 46, Section 46.111(b), including but not limited to employees (temporary, part-time, full-time, etc.) or a family member of the research staff conducting the study, or of the Sponsor, or of the Clinical Research Organization.
24. Have previously participated in a clinical trial using (Oxycodone Hydrochloride Naltrexone Hydrochloride, 1.5 mg or Oxycodone Hydrochloride , Naltrexone Hydrochloride 3.0 mg ).
25. Have a history of major mental illness that in the opinion of the Investigator may affect the ability of the subject to participate in the study. Institutionalized subjects will not be eligible for participation.
26. Been exposed to any investigational agent within 30 days or five half-lives (whichever is longer) prior to check-in for Day 1, Period 1, or is scheduled to receive an investigational device or drug (other than test product) during the course of this study.

Day -1 Exclusions:

1. Have taken any of the following drugs within the indicated times before surgery:

* over-the-counter or prescription non-steroidal anti-inflammatory drugs (NSAIDs) (such as ibuprofen [Advil®, Motrin®]), acetaminophen, or naproxen sodium (Anaprox®, Aleve®) within 24 hours; a daily dose of 81 mg of aspirin will be allowed (higher doses must be lowered to 81 mg a day by 72 hours prior to surgery).
* naproxen sodium sustained-release (Naprelan®) within 72 hours
* C-2 inhibitors (such as piroxicam or indomethacin) within 5 days
* oxycodone-containing drugs and other analgesic drugs containing opioids within the past 14 days
* immediate-release sedating antihistamines, tranquilizers, or hypnotics within at least 6 hours, or long-acting or sustained-released forms of these drugs within at least 7 days of Day -1

Day 1 Exclusion:

1. Have surgical complications (Day -1) that could compromise the safety of the subject or confound the results of the trial or any other reason that, in the opinion of the investigator, makes the subject unsuitable to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure for Oxycodone/Naltrexone (a) | Every 6 hours for 48 hours
  Self reported pain intensity prior to 1st dose, every 30 minutes for the 1st 6 hours, immediately prior to each drug administration (every 6 hours) and at 2 hours after each drug administration. Each is scored 0-10 (0=no pain and 10 = worst pain imaginable) on a Likert Scale

SECONDARY OUTCOMES:
Pain Intensity Measure for Oxycodone/Naltrexone (b) | Every 6 hours for 48 hours
  Self reported pain intensity prior to 1st dose, every 30 minutes for the 1st 6 hours, immediately prior to each drug administration (every 6 hours) and at 2 hours after each drug administration. Each is scored 0-10 (0=no pain and 10 = worst pain imaginable) on a Likert Scale
Pain Relief Measure for Oxycodone/Naltrexone (a and b formulations) | Every 6 hours for 48 hours
  Self reported pain relief, every 30 minutes for the 1st 6 hours, immediately prior to each drug administration (every 6 hours) and at 2 hours after each drug administration. Pain relief is scored on a 5 point scale of None, A Little, Some, A Lot and Complete Relief from the starting pain.
Number of Subjects with Changes in Physical Examination from Day 1 Pre-dose to End of Study | Pre-Dose Day 1 and Day 8
  Changes in Physical Exam will be evaluated/analyzed from Day 1 Pre-dose to Day 8. Descriptive statistics will be used (number and percent of occurrences).
Number of Subjects with Changes in Pulse Oximetry from Pre-Dose to post-dose time points | 48 hours (multiple time points) and at each out patient visit (Days 4, 6, 8)
  Changes in Pulse Oximetry will be evaluated/analyzed from pre-dose to post-dose values. Descriptive statistics will be used (number and present of occurrences).
Number of Subjects with Changes in Blood Chemistry Analytes from baseline to end of study | Screening, 48 hours post-dose and Day 8
  Changes in Blood Chemistry values at 48 hours post-dose and end of study will be evaluated/analyzed from baseline (screening) values. Descriptive statistics will be used (number and percent of occurrences).
Number of Subjects with Changes in Hematology Analytes from baseline to end of study | Screening, 48 hours post-dose and Day 8
  Changes in Hematology values at 48 hours post-dose and end of study will be evaluated/analyzed. Descriptive statistics will be used (number and percent of occurrences).
Number of Subjects with Changes in Urinalysis from baseline to end of study | Screening, 48 hours post-dose and Day 8
  Changes in Urinalysis at 48 hours post-dose and end of study will be evaluated/analyzed. Descriptive statistics will be used (number and percent of occurrences)
Number of Subjects with Changes in Systolic Blood Pressure from baseline through multiple post-dose time points | Pre-Dose Day 1 through Day 3, Day 4, 6, 8
  Blood pressure will be done every 6 hours for the 1st 48 hours then at each outpatient visit. Descriptive statistics will be used (number and percent of occurrences) of changes from baseline to subsequent time points post-dose.
Number of Subjects with Changes in Diastolic Blood Pressure from Baseline through multiple time points post-dose | Pre-Dose Day 1 through Day 3, Day 4, 6, 8
  Blood pressure will be done every 6 hours for the 1st 48 hours then at each outpatient visit. Descriptive statistics will be used (number and percent of occurrences) of changes from baseline to subsequent time points post-dose.
Number of Subjects with Changes in Pulse Rate | Pre-Dose Day 1 through Day 3, Day 4, 6, 8
  Pulse rate will be measured every 6 hours for the 1st 48 hours then at each outpatient visit. Descriptive statistics will be used (number and percent of occurrences) of changes from baseline to subsequent time points post-dose.
Number of Subjects with Changes in Respiratory Rate | Pre-Dose Day 1 through Day 3, Day 4, 6, 8
  Respiratory rate will be measured every 6 hours for the 1st 48 hours then at each outpatient visit. Descriptive statistics will be used (number and percent of occurrences) of changes from baseline to subsequent time points post-dose.
Number of subjects with Adverse Events as a measure of Safety and Tolerability | Day 1 through 7 days post last dose
  Number of subjects that reported an Adverse Event will be reported by body system, severity, relatedness to study drug as number and percent of occurrences.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Premier Research, Phoenix, Arizona
  - Chesapeake Research Group, Pasadena, Maryland
  - Premier Research, Austin, Texas
  - Endeavor Clinial Trials, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah